CLINICAL TRIAL: NCT06430307
Title: A Randomized, Double-blind, Placebo-controlled, Multi-center Clinical Study of Saussurea Involucrata Liquid Tonic in the Treatment of Postpartum Rheumatism
Brief Title: Efficacy and Safety of Saussurea Involucrata Liquid Tonic in Patient With Postpartum Rheumatism
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Quan Jiang (Other)
Responsible Party: Sponsor-Investigator, Quan Jiang, chief physician, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Organization: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022014P7A01
Record Dates: First submitted 2024-05-21; First posted 2024-05-28 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Postpartum Rheumatism
Keywords: Saussurea Involucrata Liquid Tonic; Traditional Chinese Medicine; Postpartum Rheumatism

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Saussurea Involucrata Liquid Tonic (Experimental): Saussurea Involucrata Liquid Tonic 20ml/time, 2 times a day, orally on an empty stomach. Total treatments 8 weeks, followed up to 12 weeks.
  Interventions: Drug: Saussurea Involucrata Liquid Tonic
- placebo of Saussurea Involucrata Liquid Tonic (Placebo Comparator): placebo of Saussurea Involucrata Liquid Tonic 20ml/time, 2 times a day, orally on an empty stomach. Total treatments 8 weeks, followed up to 12 weeks.
  Interventions: Drug: Saussurea Involucrata Liquid Tonic

INTERVENTIONS:
Drug: Saussurea Involucrata Liquid Tonic — This product is a single preparation of Saussurea Involucrata Liquid Tonic. It is used for rheumatoid arthritis, rheumatoid arthritis and dysmenorrhea caused by insufficient kidney yang and cold-damp stasis.

SUMMARY:
This study is a multi-center, randomized, double-blinded, controlled trial with two parallel arms. The study aims to evaluate the efficacy and safety of Involucrata Liquid Tonic in patients with Postpartum Rheumatism.

ELIGIBILITY:
Inclusion Criteria:

* Women experience joint and muscle pain, soreness, heaviness, numbness, etc. within 1 year after childbirth, miscarriage or induction of labor; with or without sensitivity to external stimuli such as wind, cold, moisture, etc., which may be induced or aggravated by emotional fluctuations
* Meets the diagnostic criteria for Yang Qi deficiency and cold-dampness syndrome.
* Age 18-50
* Pain VAS score ≥4cm

Exclusion Criteria:

* Those in the puerperium (within 42 days after delivery).
* Those who have rheumatoid arthritis, ankylosing spondylitis, osteitis density, polymyalgia rheumatica, reactive arthritis, myofasciitis, fibromyalgia syndrome and other rheumatic immune diseases before pregnancy.
* Severe abnormalities in blood routine and electrocardiogram, active liver disease or abnormal liver function, AST, ALT or GGT higher than 1.2 times the upper limit of normal value; abnormal renal function, serum creatinine (sCr) higher than 1.2 times the upper limit of normal value. Patients whose white blood cell count < 3.0×109/L, or hemoglobin < 90 g/L, or platelet count < 100.0×109/L in routine blood examination
* Combined with serious underlying diseases, primary diseases and postpartum diseases, such as uncontrollable hypertension, heart disease, kidney disease, puerperal fever, mastitis, moderate to severe postpartum depression diagnosed by a psychiatric department, etc.
* Those who have a history of using glucocorticoids, immunosuppressants and other drugs within 4 weeks.
* Those who are allergic to the ingredients of the test drug or have a high-sensitivity constitution.
* Existing or past history of cancer.
* Those who have participated in other clinical drug studies in the past 2 months.
* Those who do not use the medication as prescribed, or who have incomplete information that affects the judgment of efficacy.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 128 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
VAS (visual analog scale) | 8 weeks
  The number of cases with pain VAS (visual analog scale) improvement ≥30%/number of enrolled cases × 100%.

SECONDARY OUTCOMES:
SF-36 | 8 weeks
  the MOS item short from health survey, SF-36
HADS | 8 weeks
  Hospital Anxiety and Depression Scale
HAQ | 8 weeks
  Stanford Health Assessment Questionnaire
VAS | 8 weeks
  Visual Analogue Score

IPD SHARING:
Plan to Share IPD: No